CLINICAL TRIAL: NCT03588663
Title: The Acute Effect of Using a Bionic Leg on Physiological Cost Index and Biomechanical Measures in Chronic Stroke Patients
Brief Title: Effect of Using a Bionic Leg on Physiological and Biomechanical Measures in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Wright_BL_Acute_2018
Record Dates: First submitted 2018-06-11; First posted 2018-07-17 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Stroke; Physical Activity; Gait, Hemiplegic
Keywords: Robotics; Walking; Balance
MeSH Terms: conditions — Stroke; Motor Activity; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded outcomes assessor will analyse all data. Participants will not be blinded from the study as they will know whether they are using the Bionic Leg in a given testing session or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bionic Leg (Experimental): Participants will wear the Bionic Leg during a series of different activities including a timed-up-and-go, balance tests, 6-min walk test and sit-to-stand exercises.
  Interventions: Device: Baseline Bionic Leg Assessment
- Control (Active Comparator): Participants will complete a series of different activities including a timed-up-and-go, balance tests, 6-min walk test and sit-to-stand exercises without wearing the bionic leg (control condition).
  Interventions: Other: Baseline Control Condition Assessment; Other: Training; Other: Follow-up Assessment

INTERVENTIONS:
Device: Baseline Bionic Leg Assessment — The 'Bionic Leg' (BL) [Alter G, Fremont, CA, USA; approved by the Food and Drug Administration (FDA) in 2014], is an externally-wearable, battery-operated robotic device that assists patients and therapists during rehabilitation by providing adjustable and progressive functional mobility training. A patient or therapist can programme the BL to provide motor assistance during sit-to-stand exercises, over-ground walking, and stair climbing, with either more or less robotic-assistance, as desired by the therapist. As the BL increases stability and actively engages the affected leg during functional tasks, it enables patients to undertake more repetitions of specific tasks than when not wearing a BL.
  Arms: Bionic Leg
Other: Baseline Control Condition Assessment — Participants will complete identical tasks as that undertaken with the Bionic Leg, but will complete the tasks without wearing the Bionic Leg.
  Arms: Control
Other: Training — Participants will take -part in a 30-minute training session whilst wearing the Bionic Leg. The training programme will ask participants to engage in a variety of walking, balance and stair exercises. The training programme will include a 15-minute rest period after completion of the 30 minutes of exercises. This will take 45 minutes in total.
  Arms: Control
Other: Follow-up Assessment — 45 minutes after the baseline assessment, immediately following the Training programme, the following tests (PCI, TUG, postural sway, 6-min walk, sit-to-stand) will be completed. These tests will be undertaken whilst not wearing the Bionic Leg. It is anticipated that this session will last approximately 2 hours.
  Arms: Control

SUMMARY:
This study will assess the effect of wearing a wearable bionic leg, on the physiological cost index and biomechanical measures in patients with stroke. Patients will be tested during a range of activities (sit-to-stand, walking) with and without the Bionic Leg, and following a 30-min training program.

DETAILED DESCRIPTION:
The aim of this study is to investigate the acute effect of wearing a Bionic Leg on:

1. The Physiological Cost Index (PCI) and Biomechanical measures (gait, postural sway) of stroke patients compared to when they do not wear a Bionic Leg.
2. Whether after wearing a Bionic Leg for 30-minutes during a training session influences the Physiological Cost Index (PCI) and any Biomechanical measures (gait, postural sway) of stroke patients

Individuals who volunteer to participate in the present study will be asked to engage in 4 sessions in the laboratory. Firstly, participants will be asked to take part in two familiarisation sessions, which will be delivered on two separate occasions. These sessions will last one-hour each and will allow participants (stroke patients) to become accustomed to wearing and using the Bionic Leg. Sessions will consist of sit to stand, walking and stairs exercises, which will allow individuals to become familiarised with the Bionic Leg device. They will then be asked to complete 6x 10m walks to identify their self-selected walking pace. In session 3, individuals will be randomly assigned to either use the Bionic Leg, or not. Participants will initially be asked to stay seated and rested for 5 minutes so a resting heart rate can be taken. If participants are assigned to the Bionic Leg condition first, they will conduct all the following tests with the Bionic leg on, however, if not, they will perform all the tests without wearing the Bionic Leg. They will then partake in a 3-minute walk test, which will include walking at their self-selected pace (found in session 1) for 3 minutes. Following this a 15-minute rest period will be taken, and 3 x timed-up and go tests will be conducted (see outcome measures). Next, participants will be asked to take part in a balance test, and then a 6-minute walk test (see outcome measures). Following a 15-minute rest, participants will complete 10 x sit-to-stands.

During the testing session where participants are not wearing the Bionic Leg, once they have finished all of the above testing, participants will engage in further testing during this session. Following a 15-minute recovery period participants will take -part in a 30-minute training session whilst wearing the Bionic Leg. The training programme will ask participants to engage in a variety of walking, balance and stair exercises. Following this, individuals will be given a further 15-min rest period, and the original tests (PCI, TUG, postural sway, 6-min walk, sit-to-stand) which were detailed above, would be re-assessed. These tests will be undertaken whilst not wearing the Bionic Leg. It is anticipated that this session will last approximately 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of stroke within 3 months to 5 years of study start date.
* Community patients who are medically stable and are either (1) currently receiving physical therapy from a neurophysiotherapy practice or (2) attending a community-based stroke support group and do not actively receive physical therapy.
* Individuals who are able to stand and step with an aid or assistance
* Patients who are cognitively aware to undertake rehabilitation exercises, physical therapy and activity.
* Patients whose height is 1.58-1.92m
* Patients whose weight is less than 159kg.

Exclusion Criteria:

* Unresolved deep-vein thrombosis
* Unstable cardiovascular conditions
* Open wounds
* Active drug resistant infections
* Recent fractures of involved limb
* Peripheral arterial disease
* Incontinence
* Severe osteoporosis
* Non-weight bearing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Change in Physiological Cost Index between baseline and follow-up | Baseline Bionic Leg Assessment; Baseline Control Condition Assessment; Follow-up Assessment (2 hours post-baseline)
  Physiological Cost Index is a measure of energy expenditure. The Physiological Cost Index is collected from a 3-min walking test. Prior to the test, participants remain seated for 5-mins so a resting heart rate can be recorded. It is anticipated the resting heart rate will be between 40 and 80 beats per minute. Lower heart rates are considered better than higher heart rates at rest. Thereafter, participants will walk for 3 minutes at a self-selected walking pace. Heart rate will be recorded throughout. It is anticipated that the heart rate at the end of 3 minutes will be between 80 and 120 beats per minute. Lower heart rates will be seen to be better than higher heart rates. Physiological Cost Index is calculated by (Heart rate during steady state exercise - heart rate at rest)/walking speed. The smaller change in heart rate between rest and the end of the 3 minute test, the better the Physiological Cost Index.

SECONDARY OUTCOMES:
Change in Timed-Up-and-Go between baseline and follow-up | Baseline Bionic Leg Assessment; Baseline Control Condition Assessment; Follow-up Assessment (2 hours post-baseline)
  A BTS G-walk system will be used to collect Timed-Up-and-Go data. From a seated position, participants will stand, walk to a cone 3 m away, walk around the cone, and walk back to the chair and sit back down. Participants will complete 2 familiarization trials prior to the actual test itself. A minimum of 3 trials will be performed.
Change in Postural Sway between baseline and follow-up | Baseline Bionic Leg Assessment; Baseline Control Condition Assessment; Follow-up Assessment (2 hours post-baseline)
  Postural sway parameters of maximal anterior-posterior and mediolateral sway will be calculated on the basis of the center of pressure. Time series will be acquired by means of a pressure mat mounted on top of a Kistler force platform (Kistler,Winterthur, Switzerland). Participants will stand on the pressure mat, unaided if possible, and trials will consist of eyes open, shoes on; eyes closed, shoes on; eyes open, shoes off; and eyes closed, shoes off. A minimum of 3 trials will be performed for each condition, each lasting 10 s. Participants will complete this test either or with or without the Bionic Leg
Change in Gait analysis between baseline and follow-up | Baseline Bionic Leg Assessment; Baseline Control Condition Assessment; Post-Training Program Assessment
  The participants will be asked to walk for 6 m, over a pressure mat (RSscan Footscan, Ipswitch, UK), for a minimum of 3 trials in order to obtain walking gait patterns. A BTS G-Walk (Brooklyn, NewYork) sensor will also be worn by the participants to collect additional spatiotemporal gait parameters (cadence, speed, stride/step length, stance/swing phase duration, single/double support duration, and pelvic girdle angles). Participants will complete this test either or with or without the Bionic Leg
Change in 6-min walk test between baseline and follow-up | Baseline Bionic Leg Assessment; Baseline Control Condition Assessment; Follow-up Assessment (2 hours post-baseline)
  Participants will walk around two cones placed 9 m apart. Participants will walk as far as possible in 6 minutes. Participants will complete this test either or with or without the Bionic Leg.
Change in Sit-to-Stand between baseline and follow-up | Baseline Bionic Leg Assessment; Baseline Control Condition Assessment; Follow-up Assessment (2 hours post-baseline)
  10 x sit-to-stand exercises will be performed on a pressure mat

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Sport, Winchester, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no intention to share individual participant data